CLINICAL TRIAL: NCT01026207
Title: Validation of a Portable Monitoring Device for the Diagnosis of Obstructive Sleep Apnea Syndrome in Patients With Chronic Obstructive Pulmonary Disease
Brief Title: Portable Monitoring Device for the Diagnosis of Sleep Apnea in Patients With Chronic Obstructive Pulmonary Disease
Status: Terminated | Type: Observational
Why Stopped: the data was completed.
Sponsor: Associação Fundo de Incentivo à Pesquisa (Other)
Collaborators: Federal University of São Paulo (Other)
Responsible Party: Principal Investigator, Prof. Dr. Lia Azeredo-Bittencourt, Prof Dr Lia Rita Azeredo Bittencourt, Associacao Fundo de Incentivo a Psicofarmcologia
Other Study IDs: CEP1989/08
Record Dates: First submitted 2009-12-03; First posted 2009-12-04 (Estimated); Last update posted 2013-10-23 (Estimated); Status verified 2011-02

CONDITIONS: Chronic Obstructive Pulmonary Disease; Obstructive Sleep Apnea Syndrome
Keywords: Diagnostic test; polysomnography; Obstructive Sleep Apnea Syndrome; Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Sleep Apnea, Obstructive | interventions — Polysomnography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Chronic Obstructive Pulmonary Disease: Patients recruited from the Pneumology Clinic of UNIFESP, diagnosed with COPD stage II and III of Global Initiative for Chronic Obstructive Lung Disease, stable for three months, and with symptoms suggestive of Obstructive Sleep Apnea Syndrome.Patients has been underwent one night by polysomnography and one night with portable monitoring.
  Interventions: Device: Polysomnography

INTERVENTIONS:
Device: Polysomnography — Sleep study polysomnography compared with portable monitoring
  Other Names: Sleep study diagnostic

SUMMARY:
Introduction:

The prevalence of overlap between Chronic Obstructive Pulmonary Disease (COPD) and Obstructive Sleep Apnea Syndrome (OSAS) is around 10%. This overlap syndrome is an important issue because is related to nocturnal desaturation and its complications. The use of portable monitoring devices (PM) for the diagnosis of OSAS was recently accepted as an alternative to full-night polysomnography (PSG). However, there are not studies evaluating the PM recording in COPD patients to detect or exclude OSAS.

Objective:

To evaluate if a PM (Stardust®, Respironics, Inc, USA) could accurately measure the apnea-hypopnea index (AHI) in COPD patients with a suspicion of OSAS.

DETAILED DESCRIPTION:
Patients will be recruited from the Pneumology outpatient clinic of UNIFESP, Patients had been diagnosed with COPD in GOLD's stages II and III, were stable (no COPD exacerbation in the last three months), were using bronchodilators without a dose change during that period, and had symptoms suggestive of OSAS (loud snoring, reported breathing pauses during sleep and excessive sleepiness). We excluded patients with other sleep-related disorders, a diagnosis and/or previous treatment for OSAS, severe cardiovascular disorders or neuromuscular disease and those using oxygen, psychotropic drugs, alcohol or other drugs of abuse.

Patients will undergo two assessments of sleep, randomly determined: 1) PM at home for one night, 2) PM in the sleep laboratory simultaneously to the PSG. Three apnea-hypopnea index (AHI) values will be obtained and analyzed: a) AHI from PM at home, b) AHI from PM in the laboratory, and c) AHI from the PSG. Analyses of all evaluations will be performed by two trained technicians, blinded to study details.

ELIGIBILITY:
Inclusion Criteria:

* Presence of Chronic Obstructive Pulmonary Disease stage II and III of Global Initiative for Chronic Obstructive Lung Disease, stable for three months, and with symptoms suggestive of Obstructive Sleep Apnea Syndrome.

Exclusion Criteria:

* Presence of Chronic Obstructive Pulmonary Disease stage II and III

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients recruited from the Pneumology Clinic of UNIFESP, diagnosed with COPD stage II and III of Global Initiative for Chronic Obstructive Lung Disease, stable for three months, and with symptoms suggestive of Obstructive Sleep Apnea Syndrome.
Sampling Method: Probability Sample
Enrollment: 72 (Actual)
Dates: Start 2009-08; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
to evaluate the accuracy of a portable monitoring device (Stardust - STD) in the detection of patients with chronic obstructive pulmonary disease (COPD). | 2 years colect data
  compared Portable monitoring device with polysomnography in COPD patients

CONTACTS AND LOCATIONS:
Overall Officials: Lia A Bittencourt, PhD, Principal Investigator — Federal University of São Paulo
Locations (2):
- Brazil (2):
  - Associacao Fundo de Incentivo a Psicofarmacologia, São Paulo, São Paulo
  - Brazil: Associação Fundo de Incentivo à Pesquisa, São Paulo, São Paulo